CLINICAL TRIAL: NCT07052097
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase II Clinical Trial to Evaluate the Efficacy and Safety of TQC2938 Injection Combined With Background Therapy in Patients With Seasonal Allergic Rhinitis
Brief Title: Clinical Trial of TQC2938 Injection in Patients With Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQC2938-II-02
Record Dates: First submitted 2025-06-08; First posted 2025-07-04 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-04

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQC2938 injection (Experimental): TQC2938 injection, 4 weeks as a treatment cycle.
  Interventions: Drug: TQC2938 injection
- TQC2938 Placebo (Placebo Comparator): TQC2938 placebo, 4 weeks as a treatment cycle.
  Interventions: Drug: TQC2938 Placebo

INTERVENTIONS:
Drug: TQC2938 injection — TQC2938 injection is a humanized monoclonal antibody that interfering with the signal cascade.
  Arms: TQC2938 injection
Drug: TQC2938 Placebo — TQC2938 placebo, 4 weeks as a treatment cycle.
  Arms: TQC2938 Placebo

SUMMARY:
To evaluate TQC2938 injection in all patients receiving background treatment with azelastine fluticasone nasal spray. The efficacy, safety and immunogenicity of the injection in patients with seasonal allergic rhinitis compared with placebo are expected to include 136 patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 75 years at the screening period
* Patients who met the diagnostic criteria of allergic rhinitis in Chinese Guidelines for the Diagnosis and Treatment of Allergic Rhinitis (revised edition, 2022)
* Positive of at least 1 allergen skin prick test(SPT) and/or serum-specific IgE within 1 year before enrollment.
* Subjects have sufficient pollen exposure during the pollen season:
* Subjects' medical history suggested that Specific Absorption Rate (SAR) symptoms were poorly controlled or subjects' subjective symptoms were not satisfactorily controlled after drug treatment during the same pollen season in the past.
* On the day of screening, the iTNSS score in the morning was ≥6; At baseline visit, the morning iTNSS was ≥6 points, and the average score of the past 6 rTNSS was ≥6 points;
* During the screening/induction period, the subjects had good compliance;
* Subjects with asthma who were assessed by the investigator or specialist as having stable asthma;
* Voluntary participation in this trial and signing the informed consent form
* Subjects (including partners) have no pregnancy and voluntarily take one or more non-pharmaceutical measures for contraception at period from drug administration to 6 months after the last study drug administration.

Exclusion Criteria:

* Laboratory test values did not meet the requirements during screening or randomization;
* Any disease that the investigator believes interferes with the patient's ability to complete the entire course of the study;
* Patients with active autoimmune disease
* People with known or suspected immunosuppression
* Subjects with active malignancy or a history of malignancy;
* History of active pulmonary tuberculosis within 12 months prior to screening;
* Diagnosis of helminthic infection within 6 months prior to screening, not receiving standard treatment or not responding to standard treatment;
* Subjects who have undergone nasal surgery or sinus surgery within 6 months before screening
* Subjects have concomitant medical conditions that preclude them from completing the screening period assessment or evaluating the primary efficacy endpoint;
* Subjects with nasal malignancies and benign tumors;
* History of hypersensitivity to any content of the study drugs or its excipients
* Subjects with a history of systemic allergy to any biological agent;
* Pregnant or lactating women;
* Alcohol, drug and known drug dependence;
* Have a history of vital organ transplantation or hematopoietic stem cell/bone marrow transplantation;
* Any medical or psychiatric condition that, in the investigator's judgment, puts the subject at risk, interferes with participation in the study, or interferes with the interpretation of the study results;
* Any condition that the investigator or primary physician believes may not be appropriate for participating the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2025-07-31 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2025-11-28 (Actual)

PRIMARY OUTCOMES:
Retrospective nasal symptom score after 2 weeks | Baseline up to 2 weeks
  Average daily retrospective nasal symptom score (rTNSS) changed from baseline after 2 weeks of treatment. The total score is 0-12 points, with the higher score meaning the more severe symptoms.

SECONDARY OUTCOMES:
Retrospective nasal symptom score after 4 weeks | Baseline up to 4 weeks
  Mean daily retrospective nasal symptom total score (rTNSS) changes from baseline at 4 weeks of treatment. The total score is 0-12 points, with the higher score meaning the more severe symptoms.
Retrospective nasal symptom score at 2-week and 4-week at day time | Baseline up to 2 and 4 weeks
  Mean daily changes in retrospective nasal symptom total score (AM rTNSS) from baseline at 2 weeks and 4 weeks after treatment. The total score is 0-12 points, with the higher score meaning the more severe symptoms.
Retrospective nasal symptom score at 2-week and 4-week at night time | Baseline up to 2 and 4 weeks
  Mean daily nightly retrospective nasal symptom total score (PM rTNSS) changes from baseline at 2 weeks and 4 weeks after treatment. The total score is 0-12 points, with the higher score meaning the more severe symptoms.
Instantaneous nasal symptom score | Baseline up to 2 and 4 weeks
  Mean change of instantaneous nasal symptom total score (iTNSS) from baseline every morning before treatment for 2 weeks and 4 weeks. The total score is 0-12 points, with the higher score meaning the more severe symptoms.
Retrospective nasal symptom score-Mean daily rTNSS change | Baseline up to 2 and 4 weeks
  Mean daily rTNSS change from baseline at 2 weeks and 4 weeks of treatment. The total score is 0-12 points, with the higher score meaning the more severe symptoms.
Peak Inspiratory Flow | Baseline up to 2 and 4 weeks
  Mean daily changes in peak inspiratory flow from baseline at 2 weeks and 4 weeks after treatment.
Instantaneous nasal symptom score | Baseline up to 2 and 4 weeks
  Mean change rate of iTNSS from baseline before treatment at 2 weeks and 4 weeks each morning. The total score is 0-12 points, with the higher score meaning the more severe symptoms.
Instantaneous nasal single symptom score | Baseline up to 2 and 4 weeks
  Mean changes from baseline in daily retrospective nasal symptom scores (runny nose, nasal congestion, nasal itchy, and sneezing) at 2 and 4 weeks of treatment. The total score is 0-3 points, with the higher score meaning the more severe symptoms.
Instantaneous nasal single symptom score at day time | Baseline up to 2 and 4 weeks
  Mean changes from baseline in scores of individual nasal symptoms (runny nose, nasal congestion, itchy nose, and sneezing) were reviewed daily (AM) at 2 weeks and 4 weeks of treatment. The total score is 0-3 points, with the higher score meaning the more severe symptoms.
Instantaneous nasal single symptom score at night time | Baseline up to 2 and 4 weeks
  Mean changes from baseline in scores of individual nasal symptoms (runny nose, nasal congestion, nasal itchy and sneezing) at night (PM) after 2 and 4 weeks of treatment. The total score is 0-3 points, with the higher score meaning the more severe symptoms.
Retrospective ocular symptom score (rTOSS) | Baseline up to 2 and 4 weeks
  Mean changes in daily retrospective ocular symptom score (rTOSS) from baseline at 2 and 4 weeks of treatment. The total score is 0-9 points, with the higher score meaning the more severe symptoms.
Retrospective ocular symptom score (AM rTOSS) | Baseline up to 2 and 4 weeks
  Mean daily changes in retrospective ocular symptom score (AM rTOSS) from baseline at 2 weeks and 4 weeks of treatment. The total score is 0-9 points, with the higher score meaning the more severe symptoms.
Retrospective ocular symptom score (PM rTOSS) | Baseline up to 2 and 4 weeks
  Mean nightly retrospective ocular symptom score (PM rTOSS) changes from baseline at 2 weeks and 4 weeks of treatment. The total score is 0-9 points, with the higher score meaning the more severe symptoms.
Instantaneous ocular symptom score (iTOSS) | Baseline up to 2 and 4 weeks
  Mean change of instantaneous ocular symptom total score (iTOSS) from baseline every morning at 2 weeks and 4 weeks of treatment. The total score is 0-9 points, with the higher score meaning the more severe symptoms.
Retrospective ocular symptom score ( rTOSS) | Baseline up to 2 and 4 weeks
  Mean rate of change in daily rTOSS from baseline at 2 and 4 weeks of treatment. The total score is 0-9 points, with the higher score meaning the more severe symptoms.
Instantaneous ocular symptom score | Baseline up to 4 weeks
  Mean change rate of iTOSS from baseline before treatment at 2 weeks and 4 weeks each morning. The total score is 0-9 points, with the higher score meaning the more severe symptoms.
Retrospective ocular single symptom score | Baseline up to 2 and 4 weeks
  Average changes in scores of individual ocular symptoms (itchy, tearing, red eyes) at 2 and 4 weeks of treatment compared with baseline. The total score is 0-3 points, with the higher score meaning the more severe symptoms.
Retrospective ocular single symptom score | Baseline up to 2 and 4 weeks
  Average changes of individual ocular symptom scores (itchy, watery eyes, red eyes) compared with baseline were reviewed daily (AM) at 2 weeks and 4 weeks of treatment. The total score is 0-3 points, with the higher score meaning the more severe symptoms.
Retrospective ocular single symptom score | Baseline up to 2 and 4 weeks
  Average changes of individual ocular symptoms (itchy, watery eyes, red eyes) scores at night (PM) after 2 weeks of treatment and 4 weeks of treatment compared with baseline. The total score is 0-3 points, with the higher score meaning the more severe symptoms.
Quality of life questionnaire | Baseline up to 2 and 4 weeks
  Changes in quality of life questionnaire (RQLQ) scores from baseline for patients with allergic rhinitis after 2 weeks and 4 weeks of treatment. The total score is 0-168 points, with the higher score meaning the more severe symptoms.
Time of onset | Baseline up to 4 weeks
  Time of onset
Time to Reach Maximum Plasma Concentration (Tmax) | Baseline up to 4 weeks
  Curative effect peak time;
Area under the curve | Baseline up to 2 and 4 weeks
  Area under the curve of mean daily rTNSS change from baseline at 2 and 4 weeks of treatment. The total score is 0-12 points, with the higher score meaning the more severe symptoms.
Severity of nasal symptoms (e.g., Runny nose, nasal congestion, nasal itching, and sneezing.) | Baseline up to 2 and 4 weeks
  2 weeks of treatment and 4 weeks of asymptomatic or mild symptoms (e.g., Runny nose, nasal congestion, nasal itching, and sneezing.).
Adverse events and serious adverse events | Baseline up to 12 weeks
  Incidence and severity of adverse events (AE) and serious adverse events(SAE), and abnormal laboratory test indicators
Blood drug concentration | Week 0,2, 4, 8, 12 before administration
  Blood drug concentration.
Blood eosinophil (EOS) count at each evaluation visit | Week 0,2, 4, 8, 12 before administration
  Blood eosinophil (EOS) count and percentage at each evaluation visit.
Change from baseline in serum total immunoglobulin E (IgE) concentration | Week 0,2, 4, 8, 12 before administration
  Change and percentage change from baseline in serum total immunoglobulin E (IgE) concentration.
The incidence of antidrug antibodies (ADA) | Week 0,2, 4, 8, 12 before administration
  The incidence and titers of antidrug antibodies (ADA) in the test subjects. If a positive result is detected for ADA in the test subjects, then the neutralizing antibody will be tested as well.
the incidence of neutralizing antibodies (Nab) | Week 0,2, 4, 8, 12 before administration
  The incidence of neutralizing antibodies (Nab). If a positive result is detected for ADA in the test subjects, then the neutralizing antibody will be tested as well.

CONTACTS AND LOCATIONS:
Locations (30):
- China (30):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing TongRen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Ganzu Province People's Hospital, Lanzhou, Ganzu
  - Cangzhou central hosipital, Cangzhou, Hebei
  - Hebei Medical University Third Hospital, Shijiazhuang, Hebei
  - First Affiliated Hospital, Heilongjang University of Chinese Medigine, Harbin, Heilongjang
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - People'S Hospital of Zhengzhou, Zhengzhou, Henan
  - Zhengzhou Central Hospital, Zhengzhou, Henan
  - Tongji Hospital of Tongji medical college of HUST, Wuhan, Hubei
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - Northern Jiangsu People'S Hospital, Yangzhou, Jiangsu
  - The first hospital of Jilin University, Changchun, Jilin
  - China-japan Friendship Hospital, Jilin University, Changchun, Jilin
  - Affiliated Zhongshan Hospital Of Dalian university, Dalian, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University School of Medicine, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The Second People's Hospital of Shandong Province, Jinan, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Zibo Central Hospital, Zibo, Shandong
  - First Hospital of Shangxi Medical University, Taiyuan, Shangxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan